CLINICAL TRIAL: NCT03099902
Title: Association Between Maternal Smoking and GSTP1 and TNFa Polymorphism in Children With Asthma/Wheezing
Brief Title: Secondhand Smoking in Asthmatic Children
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Maria Avgeri, MD, MSc, Clinical Research Associate, AHEPA University Hospital
Other Study IDs: 14/1-3-2011
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Asthma in Children; Wheezing
Keywords: Asthma; Wheezing; GSTP1; TNFa; Secondhand smoking; Passive smoking; Intrauterine smoking
MeSH Terms: conditions — Respiratory Sounds; Asthma | interventions — Respiration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Children with asthma/wheezing whose mothers were active smokers during pregnancy
  Interventions: Diagnostic Test: Lung function; Diagnostic Test: White blood cell DNA extraction; Diagnostic Test: Urinary testing
- Controls: Children without asthma/wheezing whose mothers were active smokers during pregnancy
  Interventions: Diagnostic Test: Lung function; Diagnostic Test: White blood cell DNA extraction; Diagnostic Test: Urinary testing

INTERVENTIONS:
Diagnostic Test: Lung function — Spirometry test
Diagnostic Test: White blood cell DNA extraction — GSTP1 and TNFa polymorphisms with PCR
Diagnostic Test: Urinary testing — Urinary nicotine and cotinine detection

SUMMARY:
This study will investigate the interaction between GSTP1 / TNFa polymorphisms and passive smoking in children with asthma/wheezing. Contemporary second hand-smoke exposure will be confirmed by laboratory testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 1-18 years old with doctor diagnosed asthma/wheezing

Exclusion Criteria:

* Premature birth (< 36 gestation weeks)
* Asthma-like symptoms due to other conditions (infectious, congenital, mechanical)

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects attending the Pediatric Outpatient Clinic
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
GSTP1 and TNFa variants in children with asthma | 0 days

IPD SHARING:
Plan to Share IPD: No